CLINICAL TRIAL: NCT05109923
Title: The Effect of Onnit New Mood Supplementation in Healthy Collegiate Men and Women
Brief Title: Onnit Labs New Mood Supplementation in Healthy College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Responsible Party: Principal Investigator, Ann Brown, Assistant Professor, University of Idaho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-138
Record Dates: First submitted 2020-12-10; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Mental Health Wellness 1
Keywords: cortisol; mood

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Mood Supplementation (Experimental): The New Mood herbal supplement includes lemon balm, 5-HPT, L-Tryptophan and valerian root.
  Interventions: Dietary Supplement: Multi-Ingredient Herbal Supplement
- Placebo Supplementation (Placebo Comparator): The placebo includes rice bran and maltodextrin.
  Interventions: Dietary Supplement: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: Multi-Ingredient Herbal Supplement — Weeks 0-2 all participants consumed a placebo lead-in period and weeks 2-6 were intervention weeks. Throughout the 8 weeks (2 weeks placebo lead-in and 6 weeks intervention) participants were asked to consume 2 capsules (multi-ingredient supplement) upon waking in the morning and 2 capsules (multi-ingredient supplement) before bed.
  Arms: New Mood Supplementation
Dietary Supplement: Placebo Supplement — Weeks 0-8 all participants consumed a placebo. Throughout the 8 weeks participants were asked to consume 2 capsules (placebo) upon waking in the morning and 2 capsules (placebo) before bed.
  Arms: Placebo Supplementation

SUMMARY:
The primary purpose of this study is to assess the effectiveness of ONNIT Lab's New Mood™ dietary supplement in supporting optimal mood balance and reducing daily stress among collegiate-aged men and women. To be considered for this study, the participant must meet the following criteria: (1) current undergraduate student at the University of Idaho between 18-24 years of age, (2) have no known allergies to the ingredients of New Mood™ (Niacin, Vitamin B6, Magnesium, Valerian Extract, Lemon Balm Extract, L-Tryptophan. 5-Hydroxytryptophan, and Inositol) or the placebo (rice bran and maltodextrin), (3) not currently taking any mood/sleep supplementation or medications, (4) not currently seeking therapy or diagnosed with a psychological disorder, (5) not regularly using cigarettes, marijuana, or other illicit drugs, and (6) not pregnant or breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled collegiate men and women at the University of Idaho

Exclusion Criteria:

* Currently taking mood or sleep enhancing supplementation/medication
* Currently participating in counseling and/or therapy sessions
* Previously diagnosed with a psychological disorder

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Change in cortisol awakening response (mg/dL) over 8 weeks | Change from baseline cortisol awakening response (mg/dL) at 8 weeks
  Three salivary cortisol measurements to determine cortisol awakening response (mg/dL) from baseline to 8 weeks
Change in resting heart rate (beats per minute) over 8 weeks | Change from baseline resting heart rate (beats per minute) response at 8 weeks
  Manual radial pulse measurement of resting heart rate (beats per minute) at baseline and 8 weeks
Change in resting systolic and diastolic blood pressure (mm Hg) over 8 weeks | Change from baseline resting systolic and diastolic blood pressure (mm Hg) at 8 weeks
  Digital sphygmomanometer measurement of resting systolic and diastolic blood pressure (mm Hg) at baseline and 8 weeks
Change in depression, anxiety and stress scores (0-34) over 8 weeks | Change from baseline DASS-21 score at 8 weeks
  Depression, Anxiety and Stress Scale Questionnaire (DASS-21, 0-34) to assess depression, anxiety and stress scores from baseline to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Idaho, Moscow, Idaho, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown AF, Richardson CME, Newby N, Pulsipher S, Hoene T. Effect of a Multi-Ingredient Supplement Designed to Regulate Mood on Physiological and Psychological Outcomes: A Randomized, Double-Blind, Placebo-Controlled Trial. J Diet Suppl. 2023;20(4):631-642. doi: 10.1080/19390211.2022.2077880. Epub 2022 May 30. PMID 35635482